CLINICAL TRIAL: NCT00894751
Title: A Qualitative Comparison of Two Anesthetic Techniques in Children Undergoing Magnetic Resonance Imaging
Brief Title: Two Anesthetic Techniques in Magnetic Resonance Imaging (MRI)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low enrollment and high participant withdraw
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-0281
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Magnetic Resonance Imaging; Anesthesia
Keywords: dexmedetomidine and propofol for MRI; quality of care between two anesthetic agents for MRI
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmedetomidine (Active Comparator): Determine if there is a significant difference in the quality of care between our two standard anesthesia techniques for children undergoing a MRI of the body and/or extremity MRI.
  Interventions: Drug: dexmedetomidine
- propofol (Active Comparator): Determine if there is a significant difference in the quality of care between our two standard anesthesia techniques for children undergoing a MRI of the body and/or extremity MRI.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine general anesthesia for MRI
  Arms: dexmedetomidine
Drug: propofol — propofol general anesthesia for MRI
  Arms: propofol

SUMMARY:
The goal of this study is to determine if there is a significant difference in the quality of care between the investigators' two standard anesthesia techniques for children undergoing a MRI of the body and/or extremity MRI. Quality of care will be measured by time spent in the MRI room as well as parental satisfaction, frequency of interruptions of the MRI scan, incidence-severity of respiratory complications, post anesthesia agitation, and time spent in the induction room, MRI room, and Post-Anesthesia Care Unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting as out-patients, scheduled to receive an anesthetic for MRI of body (spine, chest, abdomen, and/or pelvis) and/or extremity (arm and/or leg).
2. The subject must be a candidate for both anesthetic techniques. This decision will be made by a staff member of the Department of Anesthesiology. This staff member will not be a member of the study team and will obtain the consent for Anesthesia.
3. The subjects must be 12 months to 7 years (inclusive of the seventh year).
4. The subject's legally authorized representative has given written informed consent to participate in the study.

Exclusion Criteria:

1. The subject is residing in the Pediatric Intensive Care Unit, the Cardiac Intensive Care Unit, or Neonatal Intensive Care Unit.
2. Anxiolytic medication is ordered before the MRI (e.g., midazolam or ketamine).
3. The subject has a history or a family (parent or sibling) history of malignant hyperthermia.
4. The subject has life-threatening, medical conditions (American Society of Anesthesiologists Physical Status 4, 5 or 6).

   * The American Society of Anesthesiologists (ASA) classification scale is a measure of physical status or how healthy the patient is.
   * For our study, we will focus on children which are defined as ASA I, II or III which means a healthy child (ASA I), a child with a systemic disease that is mild and well controlled (ASA II) or a child with systemic disease that is severe and controlled (ASA III).
5. The subject is allergic to or has a contraindication to any of the drugs used in the study.
6. The subject has previously been treated under this protocol.
7. The subject has a tracheostomy or other mechanical airway device.
8. The subject has received within the past 12 hours an oral or intravenous alpha-adrenergic, beta-adrenergic agonist, or antagonist drugs (e.g., clonidine, propranolol, albuterol).
9. The subject is not scheduled to receive anesthesia-sedation care for the MRI.
10. The subject received one of the anesthetic regimens for the same MRI during the past six months.

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be the time spent in the MRI room | 2 years

SECONDARY OUTCOMES:
Secondary outcome variables include incidence-severity of respiratory complications | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States